CLINICAL TRIAL: NCT04378881
Title: Simulation of Risk of Adverse Drug Events Associated With the Initiation of Drugs Repurposed for the Treatment of COVID-19 in Adults With Polypharmacy Using Data From Large Medicare and Commercially Insured Populations
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tabula Rasa HealthCare (Industry)
Collaborators: Cambia Health Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: COVID19-TRHC-2020-002
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: COVID; Drug Effect; Drug Interaction; Adverse Drug Event
Keywords: COVID-19; Repurposed Drug; Drug Interaction; LQTS
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study aims to perform a medication risk stratification using drug claims data and to simulate the impact of the addition of various repurposed drugs on the Medication Risk Score (MRS) in a health insurance population. Our clinical tool would enable us to identify potential multi-drug interactions and potentially reduce the risk of adverse drug events (ADE) developing in these patients infected with COVID-19.

DETAILED DESCRIPTION:
Certain investigational agents have been described in observational series or are being used anecdotally based on in vitro or extrapolated evidence. It is important to acknowledge that there are no controlled data supporting the use of any of these agents, and their efficacy for COVID-19 is unknown. FDA-approved drugs such as chloroquine/hydroxychloroquine, lopinavir/ritonavir, monoclonal IL-6 antibodies, JAK inhibitors, thalidomide, and the new investigational drug remdesivir, have been proposed for repurposing to fight COVID-19 and its complications.

A medication risk stratification strategy will be used to simulate the impacts of different potential repurposed drugs for COVID-19 and the Medication Risk Score (MRS) which is used as a predictive tool for ADEs. A retrospective study will be conducted using de-identified drug claims data for commercially insured patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled with Cambia Health Solutions; Medicare/Medicaid or Commercial Health Insurance Plan
* Patients with drug claims available from 10/01/2018 to 10/31/2019

Exclusion Criteria:

* Patients with no drug claims available for 2018
* Health Plan for injectable drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of patients will change. 95,717 patients with Medicare/Medicaid health plan and 528,436 from commercial population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-06-11 (Estimated); Study Completion 2023-11-11 (Estimated)

PRIMARY OUTCOMES:
Calculate the Medication Risk Score of de-identified participants from Medicare/Medicaid and commercial health insurance plans using their current drug regimen via our proprietary risk stratification process. | Three months
  Quantitative
Simulate the Medication Risk Score following the addition of different repurposed drugs against COVID-19 to their current drug regimen via our proprietary risk stratification process. | Three months
  Quantitative
Compare the impact (change) on the Medication Risk Score using the calculate before score and simulated after score following the addition of repurposed drugs for COVID-19 to the drug regimens of patients enrolled in the study. | Three months
  Quantitative
Measure the effects of various repurposed drugs for COVID-19 on each of the five factors computed by algorithms to derive the Medication Risk Score will be calculated via our proprietary risk stratification process. | Three months
  Quantitative

SECONDARY OUTCOMES:
Comparison of the Medication Risk Score and the effects of the addition of repurposed drugs on the drug regimen between participants with Medicare/Medicaid vs. commercial health insurance plans will be assessed. | Six months
  Qualitative
Measure the effects on Medication Risk Score of various repurposed drugs for COVID-19 within subgroups of patients classified by specific diseases or drugs used and the impact of various covariables. | One year
  Qualitative

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare Precision Pharmacotherapy Research and Development Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Application of a Novel Medication-Related Risk Stratification Strategy to a Self-Funded Employer Population. — http://www.carekinesis.com/wp-content/uploads/2018_Cicali_B_Benefits_Q_Application_of_a_novel_medication-related_risk_stratification_strategy.pdf